CLINICAL TRIAL: NCT01373437
Title: Ultrasonography in Confirming Proper Position of Endotracheal Tube in Emergency Department at Siriraj Hospital: Applicability and Accuracy
Brief Title: Ultrasonography in Confirming Proper Position of Endotracheal Tube
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Dr.Phuriphong Songarj, Department of Anesthesiology
Other Study IDs: 345/2553(EC4)
Record Dates: First submitted 2011-06-09; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Endotracheal Tube Wrongly Placed During Anesthetic Procedure
Keywords: Ultrasonography; US; Confirming; Confirmation; Proper; Position; Endotracheal tube; ETT; Emergency department; ED; Applicability; Accuracy
MeSH Terms: conditions — Emergencies | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intubate
  Interventions: Device: Ultrasonography (Sonosite )

INTERVENTIONS:
Device: Ultrasonography (Sonosite ) — Sonosite MICROMAXXTM with linear probe L38e/10-5 MHz

SUMMARY:
The purpose of this study is to assess the applicability of using ultrasonography in confirmation of the position of the endotracheal tube (ETT) after intubated to patients.

DETAILED DESCRIPTION:
To assess the applicability of using ultrasonography as compared to routine portable CXR in confirmation of ETT position.

To determine the accuracy of ultrasonography in measuring the depth of ETT as compare to standard CXR method.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old with either endotracheal or nasotracheal intubation
* having normal airway anatomy
* performed portable CXR after intubation

Exclusion Criteria:

* presence in history of neck radiation, cervical spine immobility/instability
* unstable vital signs
* unwilling to participate or denial of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who visited the emergency department, Siriraj hospital and needed ETT intubation as their adequate treatment. In the period from September 2010 to November 2010.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The confirmation of ETT depth | 1 hour
  A transcricothyroid membrane view of the ultrasonography was chosen for confirmation of ETT depth measurement. Firstly, measured the distance from probe (skin) to anterior surface of ETT. Then, measured the distance from probe (skin) to balloon cuff level. Finally the depth of ETT (Distance from vocal cord to balloon cuff) was calculated by using Pythagorus rule.

SECONDARY OUTCOMES:
The confirming the presence of ETT in airway. | 1 hour
  A transcricothyroid membrane view was chosen for confirmation of ETT position. Various glottic structures such as True Vocal Cord (TVC), False Vocal Cord (FVC), and arythenoid cartilage can be visualized.

CONTACTS AND LOCATIONS:
Overall Officials: Phuriphong Songarj, MD, Study Director — Faculty of Medicine Siriraj Hospital, Mahidol University, Thailand
Locations (1):
- Anesthesiology Department, Bangkok, Thailand